CLINICAL TRIAL: NCT05121779
Title: Head-to-head Comparison of Diagnosis Value of Pulmonary Fibrosis on 68Ga-FAPI-04 and 18F-FDG PET-CT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-NM-FAPI-PF
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — 68Ga-FAPI; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI-04 PET/CT and 18F-FDG PET/CT (Experimental): All patients diagnosed with Lung fibrosis underwent 68Ga-FAPI PET/CT and 18F-FDG PET/CT.
  Interventions: Drug: 68Ga-FAPI; Drug: 18F-FDG

INTERVENTIONS:
Drug: 68Ga-FAPI — Intravenous injection of one dosage of 18.5-22.2MBq (0.5-0.6 mCi)/Kg 68Ga-FAPI. Tracer doses of 68Ga-FAPI will be used to image lesions of pulmonary fibrosis by PET/CT.
  Other Names: 68Ga-fibroblast activating protein inhibitors
Drug: 18F-FDG — Intravenous injection of one dosage of 4.44-5.55 MBq(0.12-0.15mCi)/Kg 18F-FDG. Tracer doses of 18F-FDG will be used to image lesions of pulmonary fibrosis by PET/CT.
  Other Names: 18F-Fluorodeoxyglucose

SUMMARY:
68Ga-fibroblast activating protein inhibitors(FAPI) has been developed as a tumor-targeting agent as fibroblast activation protein is overexpressed in cancer-associated fibroblasts and some inflammation,such as inflammatory bowel disease. And it might be more sensitive than FDG in detecting a certain type of inflammations according to our preliminary research. Thus this prospective study is going to investigate whether 68Ga-FAPI PET/CT may be superior for diagnosis, therapy response assessment and follow-up of Pulmonary fibrosis than 18F-FDG PET/CT.

DETAILED DESCRIPTION:
Pulmonary fibrosis is a prototype of chronic, progressive, and fibrotic lung disease.Healthy tissue is replaced by altered extracellular matrix and alveolar architecture is destroyed, which leads to decreased lung compliance, disrupted gas exchange, and ultimately respiratory failure and death.Pulmonary fibrosis is diagnosed by identification of a pattern of usual interstitial pneumonia on the basis of radiological or histological criteria in patients without evidence of an alternative cause. Activated fibroblasts are crucial for fibrotic processes in Pulmonary fibrosis. 68Ga-FAPI has been developed as a tumortargeting agent as fibroblast activation protein is overexpressed in cancerassociated fibroblasts and inflammation. Recently，a study shows that FAPI-PET/CT imaging is a promising new imaging modality for Pulmonary fibrosis.This head-to-head comparisons aims to evaluate the severity of pulmonary fibrosis and the therapy response of 68Ga-FAPI-04 compared with 18F-FDG in the same group of pulmonary fibrosis patients.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed pulmonary fibrosis patients;
* signed written consent.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* known allergy against FAPI
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | through study completion, an average of 1 year
  Sensitivity and Specificity of 68Ga-FAPI PET/CT for Lung fibrosis in comparison with 18F-FDG PET/CT

SECONDARY OUTCOMES:
FAPI expression and SUV | through study completion, an average of 1 year
  Correlation between FAPI expression and SUV in PET
therapy response | through study completion, an average of 1 year
  Change of 68Ga-FAPI PET/CT SUVmax after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China